CLINICAL TRIAL: NCT05675943
Title: A Multicenter, Randomized, Single-blind, Placebo-controlled Clinical Study to Evaluate the Efficacy and Safety of the Anti-COVID-19 Antibody SA55 for Injection in the Treatment of Patients With Hematological Disorders Who Are Persistently Positive for the Covid-19
Brief Title: Efficacy and Safety of the Anti-COVID-19 Antibody SA55 for Injection in Patients With Hematological Disorders Who Are Persistently Positive for COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Boren Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO-SA55-0004
Record Dates: First submitted 2023-01-06; First posted 2023-01-09 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Hematological Disorders; COVID-19
Keywords: Covid-19; Hematological Disorders; Monoclonal antibody
MeSH Terms: conditions — Hematologic Diseases; COVID-19 | interventions — Injections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Anti-COVID-19 Antibody SA55 for Injection (Experimental): Anti-COVID-19 Antibody SA55 for Injection
  Interventions: Biological: Anti-COVID-19 Antibody SA55 for Injection
- Placebo (Placebo Comparator): Anti-COVID-19 Antibody SA55 for Injection administered intramuscular
  Interventions: Biological: Anti-COVID-19 Antibody SA55 for Injection

INTERVENTIONS:
Biological: Anti-COVID-19 Antibody SA55 for Injection — After the subjects are successfully screened, according to the group they belong to, they will be given the corresponding drug by intramuscular injection once (the dose of SA55 injection for subjects 40kg and above in the test group is 600mg (4ml), and the dose of SA55 injection for subjects in the test group below 40kg is 300mg (2ml), the subjects in the placebo group who are 40kg and above are injected with 4ml of placebo, and those in the test group under 40kg are injected with 2ml of placebo.The injection is allowed in both deltoid muscle of the upper arm or the buttocks muscle.

SUMMARY:
This study is a multicenter, randomized, single-blind, placebo-controlled clinical trial to evaluate the effectiveness and safety of Anti-COVID-19 Antibody SA55 for Injection in patients with hematological malignancies. This study consists of two stages. In the first stage, 8 subjects aged 18-75 were recruited for safety assessment, including the monitoring of clinical test indicators and adverse events. After confirming the preliminary safety results of the first stage, we plan to recruit 160 COVID-19 patients with hematologic disorders aged 1-75 years old and randomly divided into the SA55 group and the placebo group with a ratio of 3:1. Basic information and laboratory tests will be collected during the whole study, and the occurrence of adverse events and SAEs of all subjects were collected.

ELIGIBILITY:
Inclusion Criteria:

Subjects in this study must meet all of the following criteria:

1. Male or female patients with hematological malignancies who are in stable condition or with bone marrow failure disorders and aged from 1 to 75 years old on the day of enrollment;
2. On the day of enrollment, the subject was judged to be positive for Covid-19 nucleic acid/antigen for more than 10 days without turning negative or had turned negative but recovered positive again after 10 days;
3. On the day of enrollment, patients who have received CAR T-cell therapy, corticosteroids for a long time or other immuno-suppressive drugs, with the proportion of peripheral blood B cells is less than 2%;
4. Subjects (men and women with childbearing potential) and their sexual partners voluntarily take effective contraceptive measures from 4 weeks before screening to 3 months after the last dose of the test drug, and have no plan to donate sperm or eggs;
5. Subjects voluntarily participate in the trial and sign the informed consent form before the study begins.

Exclusion Criteria:

Those who meet any of the following conditions will be excluded:

1. Those who are known to be allergic to the test drug and any component in the preparation, or other similar drugs;
2. Complications requiring surgery within 7 days, or complication considered life-threatening within 28 days;
3. Received treatment with SARS-CoV-2 neutralizing antibody drugs before screening;
4. Convalescent plasma from recovered patients before screening;
5. Patients who took anti-SARS-CoV-2 drugs within 48 hours before enrollment, including but not limited to Paxlovid (Nirmatrelvir/Ritonavir), Azvudine, Molnupiravir, etc.
6. On the day of enrollment, meet the diagnostic criteria for severe/critical new coronavirus pneumonia;
7. Suspected to have been combined with active bacteria, fungi, viruses or other infections other than the new coronavirus;
8. Those who plan to become pregnant, are pregnant, or are breastfeeding;
9. Participated in clinical trials of SARS-CoV-2 neutralizing antibody drugs within 180 days before screening or participated in clinical trials of other drugs or medical devices within 4 weeks before screening;
10. Suffering from severe neurological diseases (epilepsy, convulsions or convulsions) or mental illness, with a family history of mental illness;
11. Suffering from other serious diseases that are not controlled, such as severe cardiovascular and cerebrovascular diseases, liver and kidney diseases, endocrine system diseases; or other diseases that the researchers judge are not suitable for participating in the study (such as currently uncontrolled autoimmune diseases, etc. );
12. Other conditions that the researcher believes are not suitable for participating in this study due to various reasons.

Ages: 1 Year to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2023-01-12 (Actual); Primary Completion 2024-04-03 (Actual); Study Completion 2024-04-03 (Actual)

PRIMARY OUTCOMES:
Time when the subject has nucleic acid and the antigen test continues to turn negative | 21 days post intramuscular injection

SECONDARY OUTCOMES:
Proportion of patients with negative persistent nucleic acid test（NAT）（key secondary endpoint） | 21 days post intramuscular injection
Change of CT value | 21 days post intramuscular injection
Proportion of Subjects Progressing to Severe/Critical | 21 days post intramuscular injection
Proportion of subjects who died from any cause | 21 days post intramuscular injection
Proportion of subjects admitted to ICU | 21 days post intramuscular injection
Number of days a case was admitted to the ICU | 21 days post intramuscular injection
Time of subject's shock correction | 21 days post intramuscular injection
Proportion of subjects requiring oxygen therapy | 21 days post intramuscular injection
Proportion of subjects requiring non-invasive ventilation | 21 days post intramuscular injection
Proportion of subjects requiring mechanical ventilation | 21 days post intramuscular injection
Days of subject's hospitalization from dosing | 21 days post intramuscular injection
Proportion of subjects with severe/critical illness or all-cause death related to COVID-19 | 21 days post intramuscular injection
The incidence of AEs | 21 days post intramuscular injection
The incidence of SAEs | 21 days post intramuscular injection

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Boren Hospital, Beijing, Beijing Municipality, China